CLINICAL TRIAL: NCT03510806
Title: Evaluation of Nutritional Supplements for Exercise Recovery
Brief Title: Nutritional Supplements for Exercise Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catherine Mikus (Industry)
Responsible Party: Sponsor-Investigator, Catherine Mikus, Senior Scientist, Beachbody
Organization: Beachbody (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 03132018BB
Record Dates: First submitted 2018-03-14; First posted 2018-04-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Post-exercise Muscle Soreness
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): taste, color, and calorie-matched to supplement
  Interventions: Other: Placebo
- Supplement (Experimental): Proprietary protein and fruit extract blend
  Interventions: Dietary Supplement: Supplement

INTERVENTIONS:
Dietary Supplement: Supplement — dietary supplement contain protein from milk and fruit extract
  Arms: Supplement
Other: Placebo — color, taste, and calorie-matched placebo
  Arms: Placebo

SUMMARY:
This study will examine the effects of nutritional supplement on post-exercise muscle soreness as well as recovery of muscle strength and function.

ELIGIBILITY:
Inclusion Criteria:

* Ability to consume supplement
* Willing to adhere to the study intervention regimen
* Willing to abstain from analgesics for duration of the study
* Agreement to adhere to Lifestyle Considerations

Exclusion Criteria:

* Current use of NSAIDs
* Use of other nutritional or herbal supplements (e.g., protein powders, tart cherry juice, BCAAs, Vitamin D, probiotics, etc.) that have been shown to effect primary or secondary outcomes
* Presence of chronic diseases, including, but not limited to, cancer, HIV, hepatitis, cardiovascular, metabolic, and orthopedic conditions
* Weight > 350 pounds
* Pregnancy or lactation
* Known food allergies or sensitivities or dietary restrictions
* Habitual consumption of > 2 alcoholic drinks per day
* Febrile illness or antibiotic use within 1 month prior to baseline testing
* Treatment with another investigational drug or other intervention within 1 month
* Current smoker or tobacco use within 1 month
* Any condition(s) or diagnosis, both physical or psychological, that, in the opinion of the principal investigator or study physician, precludes participation and/or ability to consent
* Any other factor that, in the opinion of the principal investigator or study physician, would cause harm or increased risk to the participant or close contacts, or preclude the participant's full adherence with or completion of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
post-exercise muscle soreness | 7 days
  VAS score

SECONDARY OUTCOMES:
post-exercise muscle strength | 7 days
  countermovement jump performance
post-exercise muscle function | 7 days
  repetitive countermovement jumps
satiety | 4-5 hours
  VAS scores
sleep quality | 15 days
  sleep metrics, Fitbit

CONTACTS AND LOCATIONS:
Overall Officials: Catherine R Mikus, PhD, Principal Investigator — Beachbody, LLC
Locations (1):
- Beachbody, El Segundo, California, United States

IPD SHARING:
Plan to Share IPD: Undecided